CLINICAL TRIAL: NCT05120349
Title: A Phase III, Double-blind, Randomised, Placebo-Controlled, International Study to Assess the Efficacy and Safety of Adjuvant Osimertinib Versus Placebo in Participants With EGFR Mutation-positive Stage IA2-IA3 Non-small Cell Lung Cancer, Following Complete Tumour Resection
Brief Title: A Global Study to Assess the Effects of Osimertinib in Participants With EGFRm Stage IA2-IA3 NSCLC Following Complete Tumour Resection
Acronym: ADAURA2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D516FC00001; 2023-509943-28 (Other: EU CT Number); 2021-004135-89 (EudraCT Number)
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Osimertinib; Tagrisso; NSCLC; Non-small Cell Lung Cancer; Resectable; EGFRm Positive; Adjuvant; Stage IA2-IA3
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Osimertinib (Experimental): Osimertinib 80mg, orally, once daily (Dose may be reduced to 40 mg once daily if required at the discretion of the investigator)
  Interventions: Drug: Osimertinib
- Placebo (Placebo Comparator): Matching placebo for osimertinib, orally, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Osimertinib — The initial dose of Osimertinib 80mg once daily can be reduced to 40mg once daily. Treatment can continue until disease recurrence, unacceptable toxicity or other discontinuation criteria are met.
  Other Names: AZD9291; TAGRISSO
  Arms: Osimertinib
Drug: Placebo — Matching placebo. Initial dose of 80mg once daily can be reduced to 40mg once daily.
  Arms: Placebo

SUMMARY:
This is a global study to assess the effects of osimertinib in participants with EGFRm stage IA2-IA3 non-small cell lung cancer following complete tumour resection.

DETAILED DESCRIPTION:
This is a Phase III, double-blind, randomised, placebo-controlled, 2-arm, international study assessing the efficacy and safety of adjuvant osimertinib versus placebo in participants with stage IA2-IA3 EGFRm Non-Small Cell Lung Cancer, who have previously undergone complete tumour resection. All participants must have had a tumour which harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R).

Eligible participants will be randomised in a 1:1 ratio to one of the 2 intervention arms: osimertinib 80 mg or matching placebo, once daily for 3 years unless discontinuation criteria is met.

ELIGIBILITY:
Inclusion Criteria

1. Male or female, at least ≥ 18 years.
2. NSCLC, of non-squamous histology.
3. Stage IA2 or IA3 disease, based on TNM8 classification.
4. Complete surgical resection (R0) of the primary NSCLC by lobectomy, bilobectomy, segmentectomy or sleeve resection.
5. Complete recovery from surgery at the time of randomisation. Study intervention cannot commence within 4 weeks following surgery. No more than 12 weeks may have elapsed between surgery and randomisation for participants.
6. World Health Organization performance status of 0 or 1.
7. Provision of tumour sample for central pathology assessment of pathologic risk factors and to assess EGFR mutation status prior to randomisation.
8. A tumour which harbours one of the 2 EGFR mutations (Ex19del, L858R) by cobas® EGFR Mutation Test v2 (Roche Diagnostics) or FoundationOne® test.
9. Minimum life expectancy of > 6 months.
10. Females must be using highly effective contraceptive measures, and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential. Male subjects must be willing to use barrier contraception.

Exclusion Criteria

1. Mixed small cell and non-small cell cancer history.
2. Participants with incomplete (R1/R2) resection, or who have undergone pneumonectomy or only wedge resection.
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including HCV and HIV or active uncontrolled HBV infection.
4. History of another primary malignancy, including any known or suspected synchronous primary lung cancer except for malignancy treated with curative intent with no known active disease ≥ 5 years before the first dose of study intervention and of low potential risk for recurrence.
5. Any of the following cardiac criteria:

   * Mean resting QTcF interval > 470 ms, obtained from triplicate ECGs performed at screening.
   * Any abnormalities in rhythm, conduction, or morphology of resting ECG,
   * Any factors that increase the risk of QTcF prolongation or risk of arrhythmic events.
6. History of interstitial lung disease.
7. Inadequate bone marrow reserve or organ function.
8. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study intervention.
9. Prior treatment with any anticancer therapy for NSCLC (including chemotherapy, radiotherapy, immunotherapy, and EGFR-TKIs).
10. Major surgery or significant traumatic injury within 4 weeks of the first dose of study intervention.
11. Participants currently receiving medications or herbal supplements known to be strong inducers of CYP3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2027-08-02 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) in high-risk stratum | From date of randomisation up to approximately 10 years
  DFS is defined as the time from the date of randomisation until the date of disease recurrence or date of death (by any cause in the absence of recurrence), whichever occurs first.
  Stratification to the high risk stratum will be based on pathologic features assessed by central pathology review during screening.

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) in overall population | From date of randomisation up to approximately 10 years
  DFS is defined as the time from the date of randomisation until the date of disease recurrence or date of death (by any cause in the absence of recurrence), whichever occurs first.
Overall Survival (OS) in high-risk stratum and the overall population | From date of randomization up to approximately 10 years
  OS is defined as the time from the date of randomisation until death due to any cause.
PK plasma concentrations of osimertinib and of metabolite AZ5104 in overall population | From date of randomisation up to approximately 10 years
  Ratio of metabolite-to-osimertinib to be calculated at predose, and at 0.5-2 hours postdose.
Impact of osimertinib versus placebo on physical functioning | From date of randomisation up to approximately 10 years
  Assess the impact of osimertinib versus placebo on physical functioning in both the high-risk stratum and the overall population as measured by SF-36 V2 health survey
Central Nervous System (CNS) Disease-Free Survival (DFS) in both the high-risk stratum and the overall population | From date of randomisation up to approximately 10 years
  CNS DFS is defined as the time from randomisation to the time of a CNS lesion (as assessed by investigator) or death due to any cause, regardless of whether the participant withdraws from study intervention or receives other anti-cancer therapy.
Safety and tolerability in overall population | From date of randomisation up to approximately 10 years
  AEs graded by CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Goldman, MD, Principal Investigator — University of California, Los Angeles; Yasuhiro Tsutani, MD, PhD, Principal Investigator — Kindai University Facility of Medicine; Jie He, MD, PhD, Principal Investigator — The Cancer Institute and Hospital, Chinese Academy of Medical Sciences (CAMS)
Locations (115):
- United States (14):
  - Research Site, Anchorage, Alaska
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Grand Junction, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Frederick, Maryland
  - Research Site, Morristown, New Jersey
  - Research Site, Flushing, New York
  - Research Site, New York, New York
  - Research Site, White Plains, New York
  - Research Site, Houston, Texas
  - Research Site, Fort Belvoir, Virginia
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Cipolletti
  - Research Site, La Plata
  - Research Site, Rosario
  - Research Site, S.C. de Bariloche
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Montreal, Quebec
  - Research Site, Toronto
- China (18):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Xi'an
  - Research Site, Xintai
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- Germany (6):
  - Research Site, Berlin
  - Research Site, Esslingen am Neckar
  - Research Site, Georgsmarienhütte
  - Research Site, Lübeck
  - Research Site, München
  - Research Site, Würzburg
- Italy (9):
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Roma
- Japan (13):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sakai
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Wakayama
- Malaysia (4):
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
  - Research Site, Pulau Pinang
- Poland (2):
  - Research Site, Poznan
  - Research Site, Warsaw
- Research Site, Bucharest, Romania
- Russia (2):
  - Research Site, Perm
  - Research Site, Saint Petersburg
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Málaga
  - Research Site, Valencia
  - Research Site, Vigo
  - Research Site, Zaragoza
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kadıkoy/Istanbul
- United Kingdom (5):
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Wythenshawe
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hồ Chí Minh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- See also: Lung Cancer Study Locator details (for US) — https://www.lungcancerstudylocator.com/trial/listing/310876